CLINICAL TRIAL: NCT04260243
Title: Effects of Myofascial Release in Patients with Chronic Obstructive Pulmonary Disease: a Randomized Clinical Trial
Brief Title: Myofascial Release in Patients with Chronic Obstructive Pulmonary Disease
Acronym: MFR-COPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, ARGUISUELAS MARTINEZ MARÍA DOLORES, Head of Physiotherapy, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-23
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Copd
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham Myofascial + Respiratory rehabilitation (Sham Comparator): Respiratory rehabilitation programme + sham Myofascial Release
  Interventions: Other: Sham Myofascial + Respiratory rehabilitation
- Experimental-Myofascial + Respiratory rehabilitation (Experimental): Respiratory rehabilitation programme + Myofascial Release
  Interventions: Other: Experimental-Myofascial + Respiratory rehabilitation

INTERVENTIONS:
Other: Experimental-Myofascial + Respiratory rehabilitation — 6 sessions of: Myofascial Release (20 minutes each) + Respiratory rehabilitation (60 minutes each)
  Arms: Experimental-Myofascial + Respiratory rehabilitation
Other: Sham Myofascial + Respiratory rehabilitation — 6 sessions of: Sham Myofascial Release (20 minutes each) + Respiratory rehabilitation (60 minutes each)
  Arms: Sham Myofascial + Respiratory rehabilitation

SUMMARY:
The main objective of this study is to assess the effects of a myofascial release protocol in patients with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
So far, there are no previous studies that analyze the effects of a myofascial relaxation protocol applied to the diaphragm within the respiratory rehabilitation treatment in patients with chronic obstructive pulmonary disease.

Aim: The main objective of this study is to assess the effects of a 3 weeks myofascial release protocol applied to the diaphragm on respiratory parameters in patients with chronic obstructive pulmonary disease.

Design: Randomized clinical trial

ELIGIBILITY:
Inclusion Criteria:

* COPD;
* Forced expiratory volume in the first second (FEV1) < 80%;
* FEV1/Forced vital capacity (FVC) < 70%;
* Maximal inspiratory pressure (MIP) < 70%.

Exclusion Criteria:

* Recent (6 months) spine or abdominal surgery;
* Allergic status of any kind;
* systemic diseases (rheumatic, infectious conditions, febrile state, vascular alterations, endocrine diseases including diabetes, metabolic, and neoplastic syndromes);
* neuromuscular or neurological injuries;
* previous myofascial release treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Quality of life measured with the Chronic Obstructive Pulmonary Disease Assessment Test: Score | 3 weeks
  Score (0-40) higher scores mean a worse outcome.

SECONDARY OUTCOMES:
6 Minutes Walking Test | 3 weeks
  Maximum distance reached

CONTACTS AND LOCATIONS:
Overall Officials: JUAN FRANCISCO L PÁRRAGA, Study Chair — Cardenal Herrera University

REFERENCES:
- [Background] Rocha T, Souza H, Brandao DC, Rattes C, Ribeiro L, Campos SL, Aliverti A, de Andrade AD. The Manual Diaphragm Release Technique improves diaphragmatic mobility, inspiratory capacity and exercise capacity in people with chronic obstructive pulmonary disease: a randomised trial. J Physiother. 2015 Oct;61(4):182-9. doi: 10.1016/j.jphys.2015.08.009. Epub 2015 Sep 19. PMID 26386894
- [Background] Vogelmeier CF, Criner GJ, Martinez FJ, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Chen R, Decramer M, Fabbri LM, Frith P, Halpin DM, Lopez Varela MV, Nishimura M, Roche N, Rodriguez-Roisin R, Sin DD, Singh D, Stockley R, Vestbo J, Wedzicha JA, Agusti A. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report: GOLD Executive Summary. Arch Bronconeumol. 2017 Mar;53(3):128-149. doi: 10.1016/j.arbres.2017.02.001. Epub 2017 Mar 6. English, Spanish. PMID 28274597